CLINICAL TRIAL: NCT04639817
Title: Trimethoprim-Sulfamethoxazole or Levofloxacin? A Retrospective Cohort Study of Targeted Therapy for Stenotrophomonas Maltophilia Blood Stream and Lower Respiratory Tract Infections
Brief Title: Trimethoprim-Sulfamethoxazole vs Levofloxacin as Targeted Therapy for Stenotrophomonas Maltophilia Infections: a Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: Duke University (Other); Emory University (Other)
Responsible Party: Principal Investigator, Sameer Kadri, M.D., Staff Clinician, Critical Care Medicine Department, National Institutes of Health Clinical Center (CC)
Other Study IDs: BD022382
Record Dates: First submitted 2020-11-19; First posted 2020-11-23 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Stenotrophomonas Infection
Keywords: Stenotrophomonas maltophilia, Stenotrophomonas, Levofloxacin, TMP/SMX, Trimethoprim-sulfamethoxazole
MeSH Terms: interventions — Levofloxacin; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Levofloxacin targeted therapy: Patients with Stenotrophomonas maltophilia bacteremia or lower respiratory tract infection who received Levofloxacin from day of culture positivity (day 0) through day +7.
  Interventions: Drug: Levofloxacin
- TMP/SMX targeted therapy: Patients with Stenotrophomonas maltophilia bacteremia or lower respiratory tract infection who received TMP/SMX from day of culture positivity (day 0) through day +7.
  Interventions: Drug: trimethoprim-sulfamethoxazole

INTERVENTIONS:
Drug: Levofloxacin — Levofloxacin administration
  Groups: Levofloxacin targeted therapy
Drug: trimethoprim-sulfamethoxazole — Trimethoprim-sulfamethoxazole administration
  Other Names: TMP/SMX
  Groups: TMP/SMX targeted therapy

SUMMARY:
This study seeks to compare mortality outcomes of levofloxacin and trimethoprim-sulfamethoxazole treated patients who have Stenotrophomonas maltophilia blood stream or lower respiratory tract infections by retrospectively analyzing a propensity-matched cohort from a large dataset of electronic health record data.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Stenotrophomonas maltophilia culture positive from blood or the following specified respiratory tract sites: sputum, tracheal aspirate, bronchoalveolar lavage and protected bronchial brush washings
* Received either levofloxacin or TMP/SMX targeted therapy
* Those patients that received empiric therapy with a consistent medication (for example, levofloxacin empirically in the levofloxacin targeted therapy cohort) were included

Exclusion Criteria:

* Received antimicrobial other than TMP/SMX and levofloxacin, with known activity against Stenotrophomonas maltophilia (the list of antimicrobials that fit this exclusion criteria is: erythromycin, moxifloxacin, ciprofloxacin, minocycline, tigecycline, doxycycline, eravacycline, ceftazidime, cefepime, ticarcillin-clavulanate, cefiderocol, colistin, and chloramphenicol)
* Received inconsistent empiric therapy (for example, levofloxacin empirically in the TMP/SMX targeted therapy cohort) will be excluded from analysis
* Cystic fibrosis code present
* Organism resistant to therapy received

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult inpatients with Stenotrophomonas maltophilia blood stream or lower respiratory tract infection
Sampling Method: Probability Sample
Enrollment: 1621 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Death or hospice discharge | In-hospital
  Patient died or discharged to hospice

SECONDARY OUTCOMES:
Hospital length of stay | Single encounter
  Mean hospital length of stay, where mortality will be censored as longest possible length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Kadri, MD, Principal Investigator — National Institutes of Health (NIH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
N/A, this data is deidentified

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT04639817/SAP_000.pdf